CLINICAL TRIAL: NCT05794152
Title: Wenzhou Gestational Diabetes Cohort
Acronym: WGDC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Westlake University (Other)
Collaborators: Wenzhou People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20221213ZJS001
Record Dates: First submitted 2023-02-13; First posted 2023-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes Mellitus; Intrauterine Hyperglycemia; Birth Outcome, Adverse; Nutrition, Healthy
Keywords: Precision Nutrition; Host and Microbiome; Birth Outcomes
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standardized breakfast (Other): Egg (50g), whole-wheat bread (35g), celery (30g), and dried bean curd (10g)
  Interventions: Other: Standardized breakfast
- Standardized snack (Other): Tomato (50g) and skim milk (200g)
  Interventions: Other: Standardized snack
- Standardized lunch (Other): Rice (40g), oats (40g), shrimp (70g), lettuce (80g), lean pork (30g), carrot (10g), soaked auricularia auricula (20g), broccoli (80g), cucumber (10g), tomato egg drop soup (200g), salt (3g), and oil (8g)
  Interventions: Other: Standardized lunch

INTERVENTIONS:
Other: Standardized breakfast — Participants will be provided with a standardized breakfast on a morning of the days they wear a continuous glucose monitoring (CGM) device.
  Arms: Standardized breakfast
Other: Standardized snack — Participants will be provided with a standardized snack 2 hour after they have the standardized breakfast.
  Arms: Standardized snack
Other: Standardized lunch — Participants will be provided with a standardized lunch 2 h after they have the standardized snack.
  Arms: Standardized lunch

SUMMARY:
The Wenzhou Gestational Diabetes Cohort (WGDC) is a prospective cohort study among women with gestational diabetes mellitus (GDM) during pregnancy and their offspring living in Wenzhou, China. The primary aim of this cohort is to characterize the continuous blood glucose response to dietary intake and physical activity among pregnant women with GDM over 2 weeks, and to facilitate the development of personalized nutritional/lifestyle recommendation among these patients. Another aim of the WGDC is to investigate the association of dietary and physical activity together with continuous glucose change during pregnancy on the adverse birth outcomes including preterm birth, macrosomia and large-for-gestational-age birth. The secondary aim is to investigate the prospective associations of diet, physical activity and continuous glucose change over 2 weeks among the patients with long-term metabolic health of the women and their offspring.

DETAILED DESCRIPTION:
In China, an alarming increase in the prevalence of GDM has been observed in the past decade. GDM is of concern because it is associated with several maternal and fetal medical disorders. Lifestyle changes such as diet and physical activity modifications are key for the prevention and treatment of GDM. However, the associations between dietary intake and physical activity and health outcomes for GDM women and their children remain unclear due to subjective measurements of diet and physical activity. Recently, the development of objective measurements such as food image identification and wearable activity trackers give an opportunity to gain more precise insight into these associations. In addition, for the same food and physical activity exposure, GDM women may have different blood glucose responses, but the nature of variation is currently poorly characterized. Therefore, the present WGDC design incorporates three unique components, 1) objective measurement of physical activity during pregnancy using accelerometer; 2) measurement of dietary intake using both Food Frequency Questionnaire and daily dietary records; 3) measurement of blood glucose levels over 2 weeks using continuous glucose monitors, with three standardized test meals during the 2 weeks. We will then follow up these women participants during and after this pregnancy, and also follow up their offspring.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Women with GDM mainly at 24-28 weeks of gestation
* Women intended to deliver at Wenzhou People's Hospital
* Women intended to remain in Wenzhou with their child for ≥4 years

Exclusion Criteria:

* Women with cancer and other serious medical disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2033-03-21 (Estimated)

PRIMARY OUTCOMES:
Continuous blood glucose change over 2 weeks | two weeks after enrollment
  Glucose levels are assessed by continuous glucose monitoring over 2 weeks.
Adverse birth outcomes | 9-12 weeks after enrollment
  Number of participants with adverse birth outcomes, such as, preterm birth, macrosomia and neonatal hypoglycemia.

SECONDARY OUTCOMES:
Weight changes during early childhood | at delivery, age of 6 months, 1 year, 3 years and 6 years
  Weight in kilograms
Number of participants developing type 2 diabetes | 6 years and 10 years after delivery
  Risk of developing type 2 diabetes after the delivery of the women with gestational diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (1):
- Wenzhou People's Hospital, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided